CLINICAL TRIAL: NCT02667106
Title: Systemic Pharmacokinetics of Acute, Topical, Intranasal Administration of RX0041-002 in Healthy Male and Female Subjects
Brief Title: Phase I Pharmacokinetic Study of RX0041-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmaceutical Project Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015016
Record Dates: First submitted 2016-01-18; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Drug Reaction to Analgesic Nos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-dose, open label RX0041-2 (Experimental): Active Drug
  Interventions: Drug: RX0041-2

INTERVENTIONS:
Drug: RX0041-2 — Pharmacokinetic study
  Other Names: TS

SUMMARY:
This Phase I study is to examine the systemic pharmacokinetics of RX0041-002 following acute, topical, intranasal administration to healthy male and female volunteers.

DETAILED DESCRIPTION:
This is a Phase I, single dose, single-center, open-label study of the plasma and urinary pharmacokinetics of RX004-002 and its major metabolites in male and female healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 but ≤ 80 years of age at the time of dosing.
2. BMI ≥ 18 and ≤ 32 at the screening visit.
3. Females (if of child-bearing potential and sexually active) and males (if sexually active with a partner of child-bearing potential) who agree to use a medically acceptable and effective birth control method from the first dose and for 8 days following administration of study drug. Medically acceptable methods of contraception that may be used by the participant and/or his/her partner include abstinence, birth control pills or patches, diaphragm, intrauterine device (IUD), condom, surgical sterilization, and progestin implant or injection. Prohibited methods include: the rhythm method or withdrawal.
4. Willing and able to provide written informed consent and able to understand and comply with protocol requirements.
5. During the period of study confinement, subjects will be required to abstain from beverages containing grapefruit juice or caffeine.

Exclusion Criteria:

1. Has a known allergy to any ester based anesthetics including cocaine HCl, procaine, tetracaine, chloroprocaine, dibucaine, or benzocaine Amide based anesthetic allergies are NOT exclusionary. Amide based anesthetics are: Lidocaine, mepivicaine, bupivicaine, levobupivicaine, ropivicaine, etidocaine, prilocaine, and articaine.
2. The use of amphetamines, methylphenidate or other stimulant prescription and nonprescription products such as pseudoephedrine, bronchial inhalers containing sympathomimetics (epinephrine or other beta-receptor agonist) or herbal products in the 7 days prior to screening or has a need to use these drugs during the course of the study.
3. Use of any SNRIs/SSRIs antidepressants or tricyclic antidepressant up to7 days or 5 half-lives (whichever is longer) prior to screening or has a need to use these drugs during the screening period and throughout the time period of the trial.
4. Use of MAO Inhibitor drugs up to14 days prior to screening or has a need to use these drugs during the screening period and throughout the time period of the trial.
5. Has a history of abuse of controlled substances, nasal or otherwise, or has damage to the nasal space, that in the opinion of the investigator might interfere with the ability to absorb RX0041-002.
6. Has severely traumatized mucosa or sepsis in the nasal cavity.
7. Has participated in an investigational study or received an investigational drug within 30 days preceding the randomization.
8. Is a pregnant or nursing mother.
9. Has a positive pregnancy test at Screening or Day 1.
10. Has a history of seizure, with the exception of febrile seizures.
11. Has glaucoma, symptomatic cardiovascular disease, or moderate to severe hypertension (defined as an average SBP ≥160 mmHg or an average DBP ≥ 100 mmHg at the dosing visit).
12. Has a known personal or family history of hereditary pseudocholinesterase deficiency. Study participants will be screened by asking about personal or family history of anesthetic reaction, anesthetic death, and previous diagnosis of psuedocholinesterase deficiency in a relative or personally. Subjects identified with pseudocholinesterase deficiency are at risk for delayed recovery with certain anesthetics (e.g. succinylcholine and ester-based anesthetics).
13. Has a known personal or family history of pheochromocytoma. Study participants will be specifically asked if they have been treated for a pheochromocytoma previously or if they have a family member who has been diagnosed with pheochromocytoma (since 10% of these are familial).
14. Has a known personal or family history of adrenal tumor.
15. ECG abnormalities judged clinically significant by the investigator.
16. Has a positive urine test result for drugs of abuse (amphetamines, barbiturates, cannabinoids, cocaine metabolites, opiates and oxycodone) at Screening or Day 1
17. Hematocrit, WBC, or platelets outside the normal limits and judged clinically significant by the investigator.
18. Serum potassium outside normal limits and judged clinically significant by the investigator.
19. Serum ALT, AST, and bilirubin exceeding 2X ULN for the lab's reference values.
20. Evidence of impaired renal function based upon laboratory tests and investigator opinion.
21. Clinical chemistry abnormalities judged clinically significant by the investigator.
22. Donation of blood (one pint or greater) within four weeks prior to administration of study medication.
23. Not suitable for entry into the study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Measurement of RX0041 | 24 Hours
  Cmax of RX0041
Pharmacokinetic Measurement of RX0041 | 24 Hours
  AUC of RX0041

CONTACTS AND LOCATIONS:
Overall Officials: Melissa L Goodhead, MSc, Study Director — Clinical/Regulatory Agent

IPD SHARING:
Plan to Share IPD: Undecided